CLINICAL TRIAL: NCT06473428
Title: The Association of Pulmonary Function, Diaphragm Thickness and Excursion, and Phonatory Measures in Parkinson's Disease
Brief Title: Investigating Muscle Training's Respiratory Outcomes and Voice Enhancement in Parkinson's Disease
Acronym: IMPROVE-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202306013RINA
Record Dates: First submitted 2024-05-27; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Pulmonary Disease; Voice Disorders
Keywords: Parkinson's disease; Pulmonary function; Respiratory muscle training; Diaphragm
MeSH Terms: conditions — Parkinson Disease; Lung Diseases; Voice Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory Muscle Training (Experimental): Participants in this group will undergo a specific inspiratory muscle training program. The training consists of two sessions per day, each comprising five repetitions per session. Each repetition will involve a series of inspiratory exercises aimed at strengthening the respiratory muscles. The training will be conducted six days a week for eight weeks.
  Interventions: Behavioral: respiratory muscle training
- Combined Inspiratory and Expiratory Muscle Training (Experimental): This group will participate in a combined inspiratory and expiratory muscle training regimen. Similar to the inspiratory group, training sessions will occur twice daily, with each session comprising five repetitions of both inspiratory and expiratory exercises. The training will also be conducted six days a week for eight weeks
  Interventions: Behavioral: respiratory muscle training; Behavioral: Expiratory Muscle Training
- Placebo-Controlled Expiratory Muscle Training (Placebo Comparator): Participants in this control group will receive placebo-controlled expiratory muscle training. The training sessions will be similar in structure to the experimental groups, consisting of two daily sessions with five repetitions each, conducted six days a week for eight weeks
  Interventions: Behavioral: Placebo-Controlled Expiratory Muscle Training

INTERVENTIONS:
Behavioral: respiratory muscle training — Inspiratory muscle training with two sessions per day, five repetitions per session, six days a week for eight weeks.
  Arms: Combined Inspiratory and Expiratory Muscle Training; Inspiratory Muscle Training
Behavioral: Expiratory Muscle Training — Expiratory muscle training with two sessions per day, five repetitions per session, six days a week for eight weeks.
  Arms: Combined Inspiratory and Expiratory Muscle Training
Behavioral: Placebo-Controlled Expiratory Muscle Training — Placebo-controlled expiratory muscle training with two sessions per day, five repetitions per session, six days a week for eight weeks.
  Arms: Placebo-Controlled Expiratory Muscle Training

SUMMARY:
This study aims to investigate the effects of different types of respiratory muscle training on lung function, diaphragm movement, and voice quality in patients with Parkinson's disease (PD). PD often leads to breathing difficulties and voice abnormalities due to weakened respiratory muscles and reduced diaphragm mobility. The study will involve 45 participants with PD, randomly assigned to three groups: one group will perform inspiratory muscle training, the second group will perform both inspiratory and expiratory muscle training, and the third group will receive placebo-controlled expiratory muscle training. The hypothesis is that targeted respiratory muscle training will significantly improve pulmonary function, diaphragm excursion, and phonatory measures compared to the placebo group. The findings aim to develop effective rehabilitation strategies to enhance the quality of life and communication abilities in individuals with PD.

DETAILED DESCRIPTION:
This study aims to investigate the effects of respiratory muscle training on pulmonary function, diaphragm excursion, and phonatory measures in patients with Parkinson's disease (PD). PD often leads to weakened respiratory muscles, reduced diaphragm movement, and voice abnormalities, impacting breathing and communication. The study will recruit 45 patients with PD, who will be randomly assigned to three groups: an inspiratory muscle training group, a combined inspiratory and expiratory muscle training group, and a placebo-controlled expiratory muscle training group. Over eight weeks, participants will perform daily training sessions, with the intensity of the exercises adjusted periodically. Assessments will include pulmonary function tests, ultrasound measurements of diaphragm thickness and movement, and various phonatory evaluations. The hypothesis is that respiratory muscle training will significantly improve respiratory and phonatory functions in PD patients compared to placebo, providing insights into effective rehabilitation strategies for enhancing their quality of life and communication abilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease (Hoehn & Yahr stage I-III),
* Patients aged 30-85
* Patients with stable medical condition, regular medication adherence, and ability to follow instructions.

Exclusion Criteria:

* Patients with cognitive impairment
* Patients with respiratory or other neurological diseases
* Patients with smoking history
* Patients with respiratory complications
* Patients with recent chest/abdominal surgery
* Patients with clinical instability
* Patients who are unable to perform pulmonary function tests correctly

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess the forced vital capacity (FVC) to evaluate the maximum amount of air a person can forcibly exhale from the lungs after taking the deepest breath possible.
Forced Expiratory Volume in One Second (FEV1) | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess the forced expiratory volume in one second (FEV1) to evaluate how much air a person can forcibly exhale in one second.
Maximal Inspiratory Pressure (MIP) | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess the maximal inspiratory pressure (MIP) to evaluate the strength of respiratory muscles during inhalation.
Maximal Expiratory Pressure (MEP) | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess the maximal expiratory pressure (MEP) to evaluate the strength of respiratory muscles during exhalation.
Peak Expiratory Flow Rate (PEFR) | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess the peak expiratory flow rate (PEFR) to evaluate participants' lung function.
Maximum Phonation Time | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess the maximum phonation time to evaluate the duration a participant can sustain a vowel sound.
Voice Intensity | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess voice intensity to evaluate the loudness of a participant's voice.
Speech Rate | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess speech rate to evaluate the speed at which a participant speaks.
Speech Pauses | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess speech pauses to evaluate the frequency and duration of pauses in a participant's speech.
Voice Loudness | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess voice loudness to evaluate the volume level of a participant's voice.
Voice Handicap Index (VHI-10) | Assessments will be conducted at baseline (week 0) and after the intervention period (week 8).
  This measure will assess vocal performance using the Voice Handicap Index (VHI-10) questionnaire. The VHI-10 scores range from 0 to 40, with higher scores indicating a greater perception of vocal handicap. The score interpretation is as follows: 0-10 (no or minimal handicap), 11-20 (mild handicap), 21-30 (moderate handicap), and 31-40 (severe handicap).

SECONDARY OUTCOMES:
Diaphragm Thickness | Measurements will be taken at baseline (week 0) and after the intervention period (week 8).
  This measure will assess diaphragm thickness using ultrasound to evaluate changes in diaphragm function due to the training.
Diaphragm Excursion | Measurements will be taken at baseline (week 0) and after the intervention period (week 8).
  This measure will assess diaphragm excursion using ultrasound to evaluate the movement of the diaphragm during breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-mei Yang, MD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dashtipour K, Tafreshi A, Lee J, Crawley B. Speech disorders in Parkinson's disease: pathophysiology, medical management and surgical approaches. Neurodegener Dis Manag. 2018 Oct;8(5):337-348. doi: 10.2217/nmt-2018-0021. Epub 2018 Sep 18. PMID 30223711
- [Background] Santos RBD, Fraga AS, Coriolano MDGWS, Tiburtino BF, Lins OG, Esteves ACF, Asano NMJ. Respiratory muscle strength and lung function in the stages of Parkinson's disease. J Bras Pneumol. 2019 Sep 30;45(6):e20180148. doi: 10.1590/1806-3713/e20180148. eCollection 2019. PMID 31576908
- [Background] Castillo A, Castillo J, Reyes A. Association Between Subglottic Pressure and Pulmonary Function in Individuals With Parkinson's Disease. J Voice. 2020 Sep;34(5):732-737. doi: 10.1016/j.jvoice.2019.03.001. Epub 2019 Apr 16. PMID 31000398
- [Background] Reyes A, Castillo A, Castillo J, Cornejo I. The effects of respiratory muscle training on peak cough flow in patients with Parkinson's disease: a randomized controlled study. Clin Rehabil. 2018 Oct;32(10):1317-1327. doi: 10.1177/0269215518774832. Epub 2018 May 13. PMID 29756459
- [Background] Reyes A, Castillo A, Castillo J, Cornejo I, Cruickshank T. The Effects of Respiratory Muscle Training on Phonatory Measures in Individuals with Parkinson's Disease. J Voice. 2020 Nov;34(6):894-902. doi: 10.1016/j.jvoice.2019.05.001. Epub 2019 May 31. PMID 31155431